CLINICAL TRIAL: NCT01340014
Title: Patient Preference Comparison of AZARGA Versus COSOPT in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Patient Preference Comparison of AZARGA Versus COSOPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RDG-10-251; 2010-024244-15 (EudraCT Number)
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Intraocular pressure; Tonometry, ocular
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — brinzolamide; Timolol; Azarga; dorzolamide; Ophthalmic Solutions; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZARGA/COSOPT (Other): 1 drop AZARGA instilled in each eye twice a day for 7 days, followed by 1 drop COSOPT instilled in each eye twice a day for 7 days. A 48-hour washout period separated the two treatment periods.
  Interventions: Drug: Brinzolamide 1.0% + Timolol 0.5% ophthalmic suspension; Drug: Dorzolamide 2.0% + Timolol 0.5% ophthalmic solution
- COSOPT/AZARGA (Other): 1 drop COSOPT instilled in each eye twice a day for 7 days, followed by 1 drop AZARGA instilled in each eye twice a day for 7 days. A 48-hour washout period separated the two treatment periods.
  Interventions: Drug: Brinzolamide 1.0% + Timolol 0.5% ophthalmic suspension; Drug: Dorzolamide 2.0% + Timolol 0.5% ophthalmic solution

INTERVENTIONS:
Drug: Brinzolamide 1.0% + Timolol 0.5% ophthalmic suspension
  Other Names: AZARGA®
Drug: Dorzolamide 2.0% + Timolol 0.5% ophthalmic solution
  Other Names: COSOPT®

SUMMARY:
The purpose of this study was to assess patient preference regarding ocular comfort of AZARGA® compared to COSOPT® after one week instillation of each study medication.

DETAILED DESCRIPTION:
At the Screening Visit, each intervention was instilled in one eye in a contralateral fashion to establish baseline ocular comfort prior to randomization. A 48-hour washout period separated the two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension, open-angle with or without pseudoexfoliation or pigment dispersion glaucoma in both eyes.
* On a stable regimen of intraocular pressure-lowering (IOP) medication within 30 days of Screening Visit.
* IOP considered safe (in the opinion of the Investigator) in both eyes in such a way that assures clinical stability of vision and the optic nerve throughout the study period.
* IOP between 19 and 35 millimeters mercury (mmHg) in at least one eye (study eye).
* Willing to discontinue the use of all other ocular drugs (prescribed and over-the-counter) prior to receiving the screening dose during the Screening Visit and for the entire course of the study.
* Able to follow instructions and willing and able to attend all study visits.
* Read, sign, and date an Ethics Committee reviewed and approved Informed Consent Form.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity or poor tolerance to any component of the preparations to be used in this study that is deemed clinically significant in the opinion of the Principal Investigator.
* Best corrected visual acuity worse than 20/80 Snellen in either eye.
* Any abnormality preventing reliable applanation tonometry in either eye.
* Intraocular conventional surgery or laser surgery in either eye less than 3 months prior to the Screening Visit.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the Investigator's best judgment.
* Progressive retinal or optic nerve disease from any cause.
* History of ocular herpes simplex.
* Severe allergic rhinitis or bronchial hypersensitivity that would preclude the safe administration of a topical beta-blocker.
* Bronchial asthma, a history of bronchial asthma, or severe chronic obstructive pulmonary disease that would preclude the safe administration of a topical beta-blocker.
* Women who are pregnant, lactating, or of childbearing potential and not using a reliable means of birth control.
* Participation in any other investigational study within 30 days prior to the Screening/baseline Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Severine Durier, Pharm.D, Study Director — Alcon Global Medical Affairs, Europe

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 11 study centers located in Europe.
Pre-assignment Details: This reporting group includes all enrolled participants as treated.
Groups:
- AZARGA/COSOPT: 1 drop AZARGA instilled in each eye twice a day for 7 days during Period 1, followed by 1 drop COSOPT instilled in each eye twice a day for 7 days during Period 2. A 48-hour washout period separated the two treatment periods.
- COSOPT/AZARGA: 1 drop COSOPT instilled in each eye twice a day for 7 days during Period 1, followed by 1 drop AZARGA instilled in each eye twice a day for 7 days during Period 2. A 48-hour washout period separated the two treatment periods.
Period: Period 1, First 7 Days
Arm/Group | AZARGA/COSOPT | COSOPT/AZARGA
Started | 55 | 57
Completed | 53 | 57
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Personal Reasons | 1 | 0
Period: Period 2, Second 7 Days
Arm/Group | AZARGA/COSOPT | COSOPT/AZARGA
Started | 53 | 57
Completed | 53 | 56
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all participants who completed both treatment periods and completed the preference questionnaire, per planned treatment sequence (ITT full analysis population).
Groups:
- Total: Total of all reporting groups
Arm/Group | AZARGA/COSOPT | COSOPT/AZARGA | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (10.1) | 65.0 (11.92) | 66.3 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 31 | 69
  Male | 16 | 23 | 39

OUTCOME MEASURES:

1. Primary Outcome: Preferred Treatment
Description: The participant completed a questionnaire on the Day 15 visit (ie, after administration of both study medications) consisting of a single preference question: "Thinking about the comfort of the two medications (1st and 2nd) that you took during this study, which medication do you prefer?" Preferred treatment is presented as a percentage.
Time Frame: At the end of both periods, Day 15
Population: This reporting group includes all participants who completed both treatment periods and completed the preference questionnaire, as treated.
Measure: Number; unit: Percentage of participants
Groups:
- AZARGA: 1 drop AZARGA instilled in each eye twice a day for 7 days during Period 1 or Period 2
- COSOPT: 1 drop COSOPT instilled in each eye twice a day for 7 days during Period 1 or Period 2
Arm/Group | AZARGA | COSOPT
Number analyzed (Participants) | 108 | 108
Percentage of participants | 60.2 | 39.8

2. Secondary Outcome: Ocular Discomfort
Description: Ocular discomfort was assessed by the participant 1 minute after instillation of the study medication. Ocular discomfort was rated on a 10-point scale (0=no discomfort, 9=substantial discomfort).
Time Frame: Day 7 of each period
Population: This reporting group includes all participants who completed both treatment periods and completed the preference questionnaire, as treated, minus any missing responses.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AZARGA | COSOPT
Number analyzed (Participants) | 108 | 108
Units on a scale | 2.6 (2.27) | 3.7 (2.63)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (September 2011 to October 2012). An adverse event was defined as any untoward medical condition in a subject administered a study treatment regardless of causal relationship.
Description: This reporting group includes all participants who received at least one dose of study medication. At each visit the Investigator inquired about adverse events by asking the standard question, "Have you had any health problems since your last study visit?"
Arm/Group | AZARGA | COSOPT
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/112
Other Adverse Events (participants affected / at risk) | 0/112 | 0/112

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.